CLINICAL TRIAL: NCT04368715
Title: Evaluation of Pain Perception and Wound Healing After Laser-assisted Frenectomy in Pediatric Patients: a Retrospective Comparative Study
Brief Title: Pain Perception and Wound Healing After Laser-assisted Frenectomy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, ŞİRİN GÜNER ONUR, Assist. Prof. Dr., Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUTF-BAEK 2019/481
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Frenulum; Hypertrophy
MeSH Terms: conditions — Hypertrophy | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double- blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2780 nm Er:Cr;YSGG laser treated group (Experimental): Patients treated with Er:Cr;YSGG laser for labial frenectomy
  Interventions: Device: Laser-assisted frenectomy with 2780 nm Er:Cr;YSGG and 940 nm diode laser
- 940 nm Diode laser treated group (Experimental): Patients treated with 940 nm Diode laser for labial frenectomy
  Interventions: Device: Laser-assisted frenectomy with 2780 nm Er:Cr;YSGG and 940 nm diode laser

INTERVENTIONS:
Device: Laser-assisted frenectomy with 2780 nm Er:Cr;YSGG and 940 nm diode laser

SUMMARY:
This study is based on the records of the patients treated for labial frenectomy with a dental laser at the Department of Padiatric Dentistry from January 2017 to December 2017. Patients younger than 15 years were included and in total 22 patients who matched the inclusion criteria were investigated in the study. The analyzed data included age, gender, frenelum insertion type, type of dental laser, and postoperative pain perception.

DETAILED DESCRIPTION:
This study is based on the records of the patients who received laser-assisted frenectomy treatment due to mucogingival problems at pediatric dentistry department during two year period. Twenty-two patients treated with either Er,Cr:YSGG laser 2780 nm or 940 nm diode laser were selected who fulfilled the study's inclusion criteria. The analyzed data included age, gender, frenelum insertion type, type of dental laser, postoperative pain perception and wound healing. Post-operative pain was reported with Wong-Baker Faces Pain Rating Scale after 3 hours 1, 7 and 14 days. Wound surface healing was evaluated through photography. Images were uploaded to the software and the changes in the wound area were measured in square millimeters at the day of frenectomy and on days 1, 7, and 14 postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8-13
* Patients with high frenulum insertion
* Patients without any systemic condition
* Patients treated with either treated Er:Cr;YSGG or 940 nm diode laser for labial frenectomy
* Patients who were followed up after day 1,7 and 14 for wound healing.
* Patients who were followed up after 3 hours, 1,7,14 days for pain perception

Exclusion Criteria:

* Patients with systemic condition
* Patients who were not treated with Er:Cr;YSGG or 940 nm diode laser for labial frenectomy
* Patients whose follow up was not properly completed

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Assesment of pain perception changes after laser assisted frenectomy procedure | After 3 hours, 1, 3, 7 and 14 postoperative days.
  Evaluation of changes in pain scores were evaluated with Wong-Baker Faces Pain Rating Scale which consists of a set of cartoon faces with varying facial expressions ranging from a smile/laughter to tears. Children were asked to select the facial expression that best represented their pain. Score 1 represents there is no pain, score 5 presents moderate pain and score 10 is the higher score which represents the worst pain.
Assessment of wound surface area measurement changes after laser assisted frenectomy procedure | 1, 3, 7 and 14 postoperative days.
  Evalution of wound healing. Remaining wound area (RWA): The defect area was measured after 1, 3, 7 and 14 postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: SIRIN GUNER ONUR, PhD, Study Chair — Trakya University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Onur SG. Evaluation of Pain Perception and Wound Healing After Laser-Assisted Frenectomy in Pediatric Patients: A Retrospective Comparative Study. Photobiomodul Photomed Laser Surg. 2021 Mar;39(3):204-210. doi: 10.1089/photob.2020.4886. Epub 2020 Dec 18. PMID 33337937